CLINICAL TRIAL: NCT06907121
Title: Investigation of Intra-Articular Growth Hormone and Platelet-Rich Plasma on Joint Health in Adults With Knee and Ankle Arthritis Resistant to Treatment
Brief Title: Investigation of Growth Hormone and Platelet-Rich Plasma on Joint Health
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Integrant Pty Ltd (Industry)
Collaborators: University of Technology, Sydney (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT-2025-02-12
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Arthritis Ankle; Arthritis Knee

STUDY DESIGN:
Intervention Model Description: There will be 2 groups, one with knee arthritis and one with ankle arthritis
Masking Description: Everyone receives the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment of Ankle Arthritis (Experimental): Injection of 10 iu of Somatropin and Platelet-Rich Plasma conjunct via intra-articular injection of the arthritic ankle. This will be administered with a 7-16 day buffer period between each injection. There will be three total injections for the study.
  Interventions: Drug: Intra-Articular Injection of Growth Hormone and Platelet-Rich Plasma
- Treatment of Knee Arthritis (Experimental): Injection of 10 iu of Somatropin and Platelet-Rich Plasma conjunct via intra-articular injection of the arthritic knee. This will be administered with a 7-16 day buffer period between each injection. There will be three total injections for the study.
  Interventions: Drug: Intra-Articular Injection of Growth Hormone and Platelet-Rich Plasma

INTERVENTIONS:
Drug: Intra-Articular Injection of Growth Hormone and Platelet-Rich Plasma — Intervention will be an intra-articular injection of 10 units of HGH and 10 mL PRP conjunct. Three total injections/placements of HGH spaced 7 to 16 days apart on either the effected ankle or knee joint guided by ultrasound.

SUMMARY:
This clinical study will evaluate the efficacy of intra-articular (IA) injection of growth hormone (HGH) and platelet-rich plasma (PRP) in adults with knee and ankle arthritis resistant to conventional treatment.

The study, sponsored by Integrant Pty Ltd and led by Prof. Gordon Slater, aims to determine whether IA HGH injections can enhance cartilage regeneration and joint healing.

The study will recruit 60 patients who will receive three IA injections of HGH and PRP spaced 7-16 days of each other.

Outcomes will be assessed using AOFAS and AKS scoring systems at 3- and 6-months post-treatment.

The study hypothesizes that HGH will increase healing of arthritic or injured joints compared to standard treatment, potentially providing a non-surgical alternative for patients with treatment-resistant arthritis.

DETAILED DESCRIPTION:
This clinical study will evaluate the efficacy of intra-articular (IA) injection of growth hormone (HGH) and platelet-rich plasma (PRP) in adults with knee and ankle arthritis resistant to conventional treatment. The HGH used will be approved by ethics and comes from a reputable chinese manufacturer called GenSci. The PRP Tubes are supplied by Integrant being a TGA approved device.

The study, sponsored by Integrant Pty Ltd and led by Prof. Gordon Slater, aims to determine whether IA HGH injections can enhance cartilage regeneration and joint healing. This study will be completed within Prof Gordon Slater's private clinic in a clean environment.

The study will recruit 60 patients who will receive three IA injections of HGH and PRP over 7-16 days. The inclusion criteria includes: Ankle/Knee arthritis resistant to treatment in GP clinic setting, Significant Ankle/Knee cartilage injury can be shown on MRI scan or weight bearing X-Ray within 6 months of study application, Able to give informed consent to participation in a clinical trial, Able to commit to attending clinic for follow up. The exclusion criteria include: A known hypersensitivity to any of the components of the product, Cancer diagnosis or suspicion, Resected or active tumor, Skeletally immature (<18 years of age or no radiographic evidence of closure of epiphyses), Pregnancy, Active infection at the injection site, Open soft tissue injury, Metabolic disorders known to adversely affect the skeleton (e.g. renal osteodystrophy or hypercalcemia), other than primary osteoporosis or diabetes, Over 70 years of age, Unstable joint or maligned joint > 5%, No cartilage detected in the joint (bone on bone in medical imaging), Unable to give informed consent, Unable to commit to attend clinic for follow up.

Outcomes will be assessed using AOFAS and AKS scoring systems at 3- and 6-months post-treatment. A secondary outcome of the study includes having a blood test before each injection intervention and 2 hours after each injection. This is to test for HGH within the blood of the patient.

The study hypothesizes that HGH will increase healing of arthritic or injured joints compared to standard treatment, potentially providing a non-surgical alternative for patients with treatment-resistant arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Ankle/Knee arthritis resistant to treatment in GP clinic setting.
* Significant Ankle/Knee cartilage injury can be shown on MRI scan or weight bearing X-Ray within 6 months of study application.
* Able to give informed consent to participation in a clinical trial.
* Able to commit to attending clinic for follow up.

Exclusion Criteria:

* A known hypersensitivity to any of the components of the product.
* Cancer diagnosis or suspicion.
* Resected or active tumor.
* Skeletally immature (<18 years of age or no radiographic evidence of closure of epiphyses).
* Pregnancy.
* Active infection at the injection site.
* Open soft tissue injury.
* Metabolic disorders known to adversely affect the skeleton (e.g. renal osteodystrophy or hypercalcemia), other than primary osteoporosis or diabetes.
* Over 70 years of age
* Unstable joint or maligned joint > 5%
* No cartilage detected in the joint (bone on bone in medical imaging)
* Unable to give informed consent.
* Unable to commit to attend clinic for follow up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Ankle mobility and functionality test with AOFAS scale | Baseline, 3-months after final injection, 6-months after final injection
  The AOFAS (American Orthopaedic Foot and Ankle Society) scale is a widely used outcome measure for ankle and hindfoot conditions, including ankle arthritis, assessing pain, function, and alignment, with scores ranging from 0 to 100, where higher scores indicate better function.
Knee mobility and functionality test with AKS scale | Baseline, 3-months after final injection, 6-months after final injection
  The AKS is a validated instrument used to assess patient outcomes after surgical knee interventions, evaluating both the knee joint itself (Knee Score) and functional ability (Function Score).

SECONDARY OUTCOMES:
MRI Imaging of the affected arthritic joint | Baseline, 6-months after final injection
  The MRI scans will be evaluated by a radiologist blinded to the treatment allocation to assess changes in: Cartilage volume and thickness, Synovial inflammation (e.g., synovitis), Bone marrow edema, Osteophyte formation, Other structural changes relevant to arthritis progression
Blood test for hormone | Baseline, 2 hours after each injection
  Blood tests to check for growth hormone within the blood system.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon L Slater, Professor, Principal Investigator — Integrant Pty Ltd
Locations (1):
- Dr Gordon Slater: Orthopaedic Surgeon, Potts Point, New South Wales, Australia